CLINICAL TRIAL: NCT02931864
Title: Effects of an e-Home Based Symptom Management and Mindfulness Training Programme on Quality of Life in Breast Cancer Survivors
Brief Title: Effects of an e-Home Based Symptom Management and Mindfulness Training Programme on QoL in Breast Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National University of Singapore (Other)
Collaborators: National University Hospital, Singapore (Other); National Cancer Centre, Singapore (Other)
Responsible Party: Principal Investigator, Karis Cheng, Professor, National University of Singapore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: R-545-000-073-592
Record Dates: First submitted 2016-10-10; First posted 2016-10-13 (Estimated); Last update posted 2020-09-23 (Actual); Status verified 2020-09

CONDITIONS: Breast Cancer Survivors; Symptom Management; Mindfulness Based Cognitive Therapy; Quality of Life; Oncology
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Usual care group (No Intervention): Usual care is meant the routine medical and health care services at the hospital.
- Experimental group (Experimental): Five weekly sessions of online symptom management + mindfulness training programme + usual care
  Interventions: Other: Online mindfulness training; Other: Online symptom management
- Comparison group 1 (Active Comparator): Five weekly sessions of online symptom management programme + usual care
  Interventions: Other: Online symptom management
- Comparison group 2 (Active Comparator): Five weekly sessions of online mindfulness training programme and usual care
  Interventions: Other: Online mindfulness training

INTERVENTIONS:
Other: Online mindfulness training — 5 weekly sessions of online self-administered mindfulness training programme in which they will receive audio-recorded and video-recorded instructions, pictorial or text-based instructions for various mindfulness exercises such as body scan meditation, mindful breathing and walking meditation.
  Arms: Comparison group 2; Experimental group
Other: Online symptom management — 5 weekly online education module in which they will receive video-recorded, audio-recorded, pictorial or text-based instructions for various self-management strategies. Topics include fatigue, pain, numbness/tingling, lymphedema, anxiety/depression, and problems with sleeping.
  Arms: Comparison group 1; Experimental group

SUMMARY:
Breast cancer is the most common cancer in women in Singapore. Breast cancer survivors usually experience side effects/symptoms after surgery and/or adjuvant chemotherapy and/or radiotherapy such as fatigue, lymphedema, problems with sleeping, peripheral neuropathy, and anxiety/depression. Currently, there is no study to include both symptom management and mindfulness training components for breast cancer survivors. And given breast cancer survivors have infrequent clinical follow-up, we aim to develop an e-Home based symptom management and mindfulness training programme for breast cancer survivors and to determine its effects on quality of life, symptom distress, psychosocial adjustment, psychological morbidity, and unplanned outpatient attendance or hospitalisation in breast cancer survivors. We employ a randomised clinical trial with four study arms (with 47 subjects in each arm) together with a process evaluation; group 1 (usual care), group 2 (experimental group: five weekly sessions of online symptom management + mindfulness training programme and usual care), group 3 (comparison group 1: five weekly sessions of online symptom management programme and usual care), and group 4 (comparison group 2: five weekly sessions of online mindfulness training programme and usual care). Subjects will complete questionnaires measures of 6-item Social Support Questionnaire, Breast Cancer Survivor Self-Efficacy Scale, the Quality of Life-Cancer Survivor Scale, Memorial Symptom Assessment Scale, Psychosocial Adjustment to Illness Scale, short version of the Fear of Recurrence Scale, Hospital and anxiety Depression Scale and Five Facet Mindfulness Questionnaire at baseline (printed questionnaires), at 8 weeks from baseline, at 12 weeks from baseline and at 24 weeks from baseline by an online system or printed questionnaires. Individualised semi-structured interview (15-25 mins) for experimental and comparison groups will be conducted at 24 weeks from baseline to understand the subjects' experiences of the study programme. Data will be analysed using SPSS version 24. Baseline demographic and clinical information of subjects in the experimental, comparison and control groups will be summarised using descriptive statistics, and will be compared using chi square tests and ANOVA/ANCOVA tests. Intention-to-treat approach will be used. Repeated measures analysis of variance will be used to examine the differences on outcome measures among the experimental, comparison and control groups across study time points. In addition, differences in changes in outcome measures among experimental, comparison groups and usual care groups will be tested using multilevel modelling techniques. A p-value smaller than 5% will be considered as statistically significant. Content analysis will be conducted to analyse the interviews data.

ELIGIBILITY:
Inclusion Criteria:

* women aged 21 or above
* able to speak and read English
* diagnosed with breast cancer stage 0 to 3 for the first time
* have completed cancer treatment including breast surgery and/or adjuvant chemotherapy and/or radiotherapy between 6 months to 5 years previously
* with and without ongoing HER2 target therapy (e.g.: Herceptin) and/or hormonal therapy
* with ECOG Performance Status score of 0 to 1
* able to understand the study and give informed consent
* have access to the internet through a handheld device

Exclusion Criteria:

* they are illiterate
* have serious psychiatric disorders (e.g. schizophrenia, dementia, and intellectual disabilities)
* with ECOG Performance Status score of 2 or above

Ages: 21 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 172 (Actual)
Dates: Start 2016-12-06 (Actual); Primary Completion 2020-03-14 (Actual); Study Completion 2020-03-14 (Actual)

PRIMARY OUTCOMES:
Change from baseline quality of life score at 8 weeks | Change between baseline and at 8 weeks
Change from baseline quality of life score at 12 weeks | Change between baseline and at 12 weeks
Change from baseline quality of life score at 24 weeks | Change between baseline and at 24 weeks

SECONDARY OUTCOMES:
Change from baseline social support score at 8 weeks | Change between baseline and at 8 weeks
Change from baseline social support score at 12 weeks | Change between baseline and at 12 weeks
Change from baseline social support score at 24 weeks | Change between baseline and at 24 weeks
Change from baseline self-efficacy score at 8 weeks | Change between baseline and at 8 weeks
Change from baseline self-efficacy score at 12 weeks | Change between baseline and at 12 weeks
Change from baseline self-efficacy score at 24 weeks | Change between baseline and at 24 weeks
Change from baseline symptom score at 8 weeks | Change between baseline and at 8 weeks
Change from baseline symptom score at 12 weeks | Change between baseline and at 12 weeks
Change from baseline symptom score at 24 weeks | Change between baseline and at 24 weeks
Change from baseline psychosocial adjustment to illness score at 8 weeks | Change between baseline and at 8 weeks
Change from baseline psychosocial adjustment to illness score at 12 weeks | Change between baseline and at 12 weeks
Change from baseline psychosocial adjustment to illness score at 24 weeks | Change between baseline and at 24 weeks
Change from baseline fear of recurrence score at 8 weeks | Change between baseline and at 8 weeks
Change from baseline fear of recurrence score at 12 weeks | Change between baseline and at 12 weeks
Change from baseline fear of recurrence score at 24 weeks | Change between baseline and at 24 weeks
Change from baseline anxiety and depression score at 8 weeks | Change between baseline and at 8 weeks
Change from baseline anxiety and depression score at 12 weeks | Change between baseline and at 12 weeks
Change from baseline anxiety and depression score at 24 weeks | Change between baseline and at 24 weeks
Change from baseline mindfulness score at 8 weeks | Change between baseline and at 8 weeks
Change from baseline mindfulness score at 12 weeks | Change between baseline and at 12 weeks
Change from baseline mindfulness score at 24 weeks | Change between baseline and at 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Karis Cheng, Principal Investigator — National University of Singapore
Locations (2):
- Singapore (2):
  - National Cancer Centre Singapore, Singapore
  - National University Hospital, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cheng KK, Darshini Devi R, Wong WH, Koh C. Perceived symptoms and the supportive care needs of breast cancer survivors six months to five years post-treatment period. Eur J Oncol Nurs. 2014 Feb;18(1):3-9. doi: 10.1016/j.ejon.2013.10.005. Epub 2013 Dec 5. PMID 24315730
- [Background] Ferrell BR, Dow KH, Grant M. Measurement of the quality of life in cancer survivors. Qual Life Res. 1995 Dec;4(6):523-31. doi: 10.1007/BF00634747. PMID 8556012
- [Background] Portenoy RK, Thaler HT, Kornblith AB, Lepore JM, Friedlander-Klar H, Kiyasu E, Sobel K, Coyle N, Kemeny N, Norton L, et al. The Memorial Symptom Assessment Scale: an instrument for the evaluation of symptom prevalence, characteristics and distress. Eur J Cancer. 1994;30A(9):1326-36. doi: 10.1016/0959-8049(94)90182-1. PMID 7999421
- [Background] Bower JE, Ganz PA, Desmond KA, Bernaards C, Rowland JH, Meyerowitz BE, Belin TR. Fatigue in long-term breast carcinoma survivors: a longitudinal investigation. Cancer. 2006 Feb 15;106(4):751-8. doi: 10.1002/cncr.21671. PMID 16400678
- [Background] Zigmond AS, Snaith RP. The hospital anxiety and depression scale. Acta Psychiatr Scand. 1983 Jun;67(6):361-70. doi: 10.1111/j.1600-0447.1983.tb09716.x. PMID 6880820
- [Background] Baer RA, Smith GT, Hopkins J, Krietemeyer J, Toney L. Using self-report assessment methods to explore facets of mindfulness. Assessment. 2006 Mar;13(1):27-45. doi: 10.1177/1073191105283504. PMID 16443717
- [Background] Champion VL, Ziner KW, Monahan PO, Stump TE, Cella D, Smith LG, Bell CJ, Von Ah D, Sledge GW. Development and psychometric testing of a breast cancer survivor self-efficacy scale. Oncol Nurs Forum. 2013 Nov;40(6):E403-10. doi: 10.1188/13.ONF.E403-E410. PMID 24161644